CLINICAL TRIAL: NCT03174678
Title: The Effect of Oral Dexmedetomidine Premedication On Preoperative Cooperation and Emergence Delirium In Children Undergoing Dental Treatment
Brief Title: Dexmedetomidine Premedication in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SULTAN KELES, Assist. Prof.Dr., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017/1080
Record Dates: First submitted 2017-05-28; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Premedication
Keywords: Dexmedetomidine; child; premedication; emergence delirium; dental treatment
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Retrospective study
Who Masked: Investigator
Masking Description: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine (Experimental): Group administered 1µg/kg dexmedetomidine oral
  Interventions: Drug: Dexmedetomidine
- Control (Other): Apple juice
  Interventions: Other: apple juice

INTERVENTIONS:
Drug: Dexmedetomidine — 1µg/kg dexmedetomidine oral
  Other Names: Precedex
  Arms: Dexmedetomidine
Other: apple juice — apple juice
  Arms: Control

SUMMARY:
The aim of this retrospective study was to detect the effectiveness of 1µg/kg oral dexmedetomidine premedication on preoperative cooperation and emergence delirium of the the young children underwent complete dental treatment.

DETAILED DESCRIPTION:
One Hundred children between the ages 2-6 years of ASA I status underwent full mouth dental rehabilitation were enrolled in the study. Group Dex (n=50) received 1µg/kg dexmedetomidine in apple juice and Group control (n=50) received apple juice only. Patients' Ramsey Sedation Scale (RSS), The Parental Seperation Anxiety Scale (PSAS), Mask Acceptance Scale (MAS) and Post anesthesia emergence delirium scale (PAEDS) and hemodynamic parameters were noted from their patient file. Premedication period was 45 minutes and measurements of RSS and hemodynamic parameters were recorded in baseline and every 15 minutes until the patients were transferred to the operating room. The data were analysed using the Kruskal-Wallis test, two sample t- tests, chi-square tests and ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria is age between 2 to 6 years and American Society og Anesthesiology (ASA) grade 1.

Exclusion Criteria:

* The exclusion criteria included congenital disease, DEX, propofol allergy, asthma, mental retardation and those children parents refuse to participate study.

Ages: 2 Years to 6 Years | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Ramsey Sedation Score | 45 minutes after premedication
  Sedation level

SECONDARY OUTCOMES:
Parental Separation Anxiety Score | preoperative
  Separation anxiety

OTHER OUTCOMES:
Mask Acceptance Score | Before induction
  Mask acceptance

CONTACTS AND LOCATIONS:
Overall Officials: sultan keles, Dr., Principal Investigator — Pediatric dentistry
Locations (1):
- Sultan Keles, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kumari S, Agrawal N, Usha G, Talwar V, Gupta P. Comparison of Oral Clonidine, Oral Dexmedetomidine, and Oral Midazolam for Premedication in Pediatric Patients Undergoing Elective Surgery. Anesth Essays Res. 2017 Jan-Mar;11(1):185-191. doi: 10.4103/0259-1162.194586. PMID 28298782
- [Derived] Keles S, Kocaturk O. The Effect of Oral Dexmedetomidine Premedication on Preoperative Cooperation and Emergence Delirium in Children Undergoing Dental Procedures. Biomed Res Int. 2017;2017:6742183. doi: 10.1155/2017/6742183. Epub 2017 Aug 20. PMID 28904966